CLINICAL TRIAL: NCT06665828
Title: A Phase 1, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of REGN9533, a Monoclonal Antibody Against Factor XII, in Healthy Adults
Brief Title: Phase 1 Safety and Tolerability Study of REGN9533 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R9533-HV-2411; 2024-515285-14-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- REGN9533 (Experimental): Randomized as described in the protocol Escalating Cohorts including Optional Cohorts
  Interventions: Drug: REGN9533
- Placebo (Experimental): Randomized as described in the protocol
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: REGN9533 — Administered per the protocol
  Arms: REGN9533
Drug: Matching Placebo — Administered per the protocol.
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to see how safe and tolerable the clinical trial drug (REGN9533) is in healthy participants. This is the first time that REGN9533 will be given to humans.

After the clinical trial drug has been tested in healthy participants, future studies with REGN9533 will focus on participants with thromboembolic (blocking of blood vessels) diseases which include blood clots.

REGN9533 is a drug that is only used in clinical studies.

The clinical trial is looking at:

* The side effects REGN9533 might cause
* How much REGN9533 is in the blood at different times
* How the body reacts to REGN9533
* If the body makes antibodies to REGN9533 (unwanted immune response, which may cause REGN9533 to not work as well)
* What is the best dose of REGN9533

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a body mass index between 18 and 32 kg/m2, inclusive
2. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and electrocardiograms (ECGs) performed at screening and/or prior to administration of initial dose of study drug
3. Normal aPTT, normal PT, and normal platelet counts as described in the protocol
4. Hemoglobin values at screening period and at day -1 as described in the protocol
5. Negative Fecal Occult Blood Test (FOBT) during screening period
6. Normal Bleeding Time Test (BTT) at day -1 as defined by the study site

Key Exclusion Criteria:

1. History of any major surgical procedure or clinically significant physical trauma within the last 6 months that in the opinion of the investigator may pose a risk to the participant by study participation
2. History of clinically significant bleeding, requiring hospitalization or blood products within the last 6 months, that in the opinion of the investigator may pose a risk to the participant by study participation
3. History of bleeding diathesis (eg, including, but not limited to Hemophilia A or B, von Willebrand's Factor deficiency, fibrinogen deficiency, and other inherited or acquired bleeding disorders)
4. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease, as assessed by the investigator, that may confound the results of the study or poses an additional risk to the participant by study participation
5. Is a current smoker including e-cigarettes or other nicotine-containing products; or is a former smoker including e-cigarettes or other nicotine-containing products which they have used at any time within 3 months prior to the screening visit
6. Has a confirmed positive drug test result at the screening visit and/or prior to randomization; or a history of recreational drug use (eg, marijuana) and/or drug or alcohol abuse within a year prior to the screening visit
7. Any malignancy, except for non-melanoma skin cancer or cervical/anus in-situ, that have been resected with no evidence of metastatic disease for 3 years prior to the screening visit
8. Has a history of significant multiple and/or severe allergies (eg, latex gloves), or has had an anaphylactic reaction to prescription or non-prescription drugs or food

Note: Other protocol-defined Inclusion/Exclusion Criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-01-29 (Actual); Study Completion 2026-01-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Up to 100 days
Severity of TEAEs | Up to 100 days

SECONDARY OUTCOMES:
Change in activated Partial Thromboplastin Time (aPTT) | Baseline up to 100 days
Change in Prothrombin Time (PT) | Baseline up to 100 days
Concentrations of REGN9533 | Up to 100 days
Incidence of Anti-drug Antibodies (ADAs) to REGN9533 | Up to 100 days
Titer of ADAs to REGN9533 | Up to 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- SGS Belgium NV_Edegem, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/